CLINICAL TRIAL: NCT02345746
Title: Phase 2 Study of Hepatic Arterial Infusion With Oxaliplatin, Folinic Acid and 5 Fluorouracil Alone or in Combination With Intravenous Chemotherapy in Heavily Pre-Treated Patients With Liver-Predominant Metastasis From Colorectal Cancer
Brief Title: Hepatic Arterial Infusion With FOLFOX Alone or in Combination With IV Chemotherapy in Colon Cancer With Liver Metastasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: patient population
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Principal Investigator, Jordan Waypa, Research Director, Western Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-19
Record Dates: First submitted 2013-06-12; First posted 2015-01-26 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hepatic Artery Infusion (Experimental): Hepatic Arterial Infusion (HAI) with the drugs Oxaliplatin, Folinic Acid and 5 Fluorouracil
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin — infusion over 12 hours via HAI
  Other Names: Eloxatin®
Drug: Folinic Acid — as a 2-hour infusion via HAI on day 2
  Other Names: Leucovorin
Drug: 5-Fluorouracil — Following Folinic Acid as a continuous infusion over 48 hours on days 2, 3
  Other Names: 5-FU

SUMMARY:
In this study, Hepatic Arterial Infusion will be combined with systemic therapy for patients with liver-only or liver-predominant metastases who have failed at least one line of systemic chemotherapy.

DETAILED DESCRIPTION:
In this phase II study, investigators will combine the HAI with systemic therapy for patients with liver-only or liver-predominant metastases who have failed at least one line of systemic chemotherapy. We hypothesize that combination therapy will be able to convert some patients to surgical resection candidates, or/and to overcome chemo-resistance of liver metastases to systemic i.v. chemotherapy for some clinically fit, heavily pre-treated patients

ELIGIBILITY:
Inclusion Criteria:

1. Performance status ECOG 0-2 and a life expectancy of >3 months.
2. Patients were required to have measurable disease in the liver, defined as lesions measuring >1 cm in largest diameter on spiral-computed tomography (CT) or magnetic resonance imaging (MRI)
3. Histologically confirmed metastatic advanced solid tumors involving the liver, liver replacement less than 70%
4. No bevacizumab (avastin) use within 4 weeks prior to enrollment.
5. Absence of portal vein thrombosis
6. Not a surgical candidate or patients refuse surgery
7. Loss of response to at least two lines of systemic chemotherapy including FU, Oxaliplatin or irinotecan in metastatic setting
8. An asymptomatic extra-hepatic disease is allowed, provided that the extent of the metastatic disease in the liver represented the bulk of the metastatic disease.
9. History of liver-directed therapy is eligible at the investigator's discretion.
10. Adequate renal function with a calculated creatinine clearance greater than 60 mL/min.
11. Hepatic function as follows: Total Bilirubin ≤3 mg/dL, AST ≤5 times upper normal reference value, or ALT ≤ 5 times upper normal reference value.
12. Adequate bone marrow function (ANC ≥1500 cells/uL; PLT ≥ 100,000 cells/uL) before each therapy.
13. At least three weeks from previous immunotherapy, chemotherapy or radiotherapy before being enrolled in this study.
14. All females in childbearing age MUST have a negative serum HCG test unless patients have prior hysterectomy. Women of childbearing potential must take adequate precautions to prevent pregnancy during treatment.
15. Patient consent must be obtained prior to entrance onto study

Exclusion Criteria:

1. Clinical or radiographic evidence of moderate amount of ascites.
2. History of cirrhosis with Child-Pugh class B or C.
3. Pregnant or lactating females.
4. Inability to complete informed consent process and adhere to protocol treatment plan and follow-up requirements.
5. Patients receiving any other investigational agents.
6. Patients with bleeding diathesis (clinical bleeding, prothrombin time =/> 1.5 X upper institutional normal value, INR =/> 1.5, activated partial thromboplastin time aPTT =/> 1.5 X upper institutional normal value), active gastric or duodenal ulcer.
7. History of thrombophilia, recurrent DVTs, diagnosis of phospholipid syndrome.
8. Past or current history of malignancy other than colon cancer with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a DFS ≥5 years.
9. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.
10. Patients with clinically significant cardiovascular disease: myocardial infarction or unstable angina within 6 months, New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris, clinically significant peripheral vascular disease
11. Patients have untreated brain metastasis or leptomeningeal metastases requiring immediate intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Determine response rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jiaxin Niu, MD, Principal Investigator — Western Regional Medical Center